CLINICAL TRIAL: NCT04926376
Title: Investigation of Safety and Effectiveness of Eye90 Microspheres™ in the Treatment of Unresectable Hepatocellular Carcinoma (HCC) and Metastatic Colorectal Cancer (mCRC)
Brief Title: Safety and Effectiveness of Eye90 Microspheres™ in the Treatment of Unresectable Hepatocellular Carcinoma (HCC) and Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABK Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABK-QA-PROT-37
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Metastatic Colorectal Cancer; Liver Cancer
Keywords: Hepatocellular Carcinoma; Metastatic Colorectal Cancer; Liver Neoplasms; Liver Diseases; Internal radiation brachytherapy; Radioembolization; Y90; Yttrium-90; Eye90 microspheres
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- EYE90 Microspheres Treament (Experimental): Radioembolization with Eye90 Microspheres
  Interventions: Device: Eye90 Microspheres

INTERVENTIONS:
Device: Eye90 Microspheres — Y90 glass microspheres

SUMMARY:
The purpose of this study is to evaluate the safety of treatment with Eye90 microspheres in patients with unresectable Hepatocellular Carcinoma (HCC) and metastatic Colorectal Cancer (mCRC). Both cause tumors, known as malignant hyper-vascular hepatic neoplasia, that have an abnormally large number of blood vessels attached to them. Eye90 is internal radiation brachytherapy for treatment of malignant hyper-vascular hepatic neoplasia that uses microspheres, tiny glass beads smaller in diameter than a human hair, to provide radiation. The microspheres contain Yttrium-90 (Y90) as the radiation source, which are used to to kill cancer cells and shrink tumors. The microspheres are also radiopaque, which means that they can be seen during imaging procedures. The visibility of the microspheres allows the study doctor to confirm the microspheres have been delivered in the tumor; this may help to improve the outcome of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease defined as at least one unidimensional measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI).
* Must have at least one lesion > 2 cm within the target perfused volume.
* At least one lesion must meet the definition of target lesion as defined by RECIST 1.1 or mRECIST.
* Total linear length of all lesions must be ≤ 9 cm.
* Must have preservation of >700cc of normal liver parenchyma outside of treated volume.
* Hypervascular lesions on CT scan with 99mTC MAA SPECT/CT T:N ratio 3:1 or higher and Hypervascular on CBCT.
* No prior locoregional therapies in the liver other than previous Drug Eluting Bead TACE and/or local HCC recurrence after thermal ablation. Last TACE and/or ablation treatment must be at least 3 months prior to informed consent. Prior Lumi or Lipiodol TACE is not allowed.
* Life expectancy of ≥ 6 months.
* ≥ 18 years old.

Exclusion Criteria:

* Hemoglobin ≤ 85 mg/L.
* Platelet count < 50,000/microliter or prothrombin (PT) activity > 50% normal
* INR > 1.4 (if anticoagulated, reversal must be achieved prior to any angiographic procedures).
* ALT > 2.5x upper limit
* AST > 2.5x upper limit
* For HCC subjects, Bilirubin ≥ 2 mg/dL.
* For mCRC subjects, Bilirubin ≥ 1.2 mg/dL.
* eGFR ≤ 60 mL/min/1.73 m2.
* Portal vein thrombosis (PVT).
* Incompetent biliary duct system, prior biliary intervention, or a compromised Ampulla of Vater
* Estimated lung dose > 30 Gy as calculated using the lung shunt % and partition model.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | 6 months
  Incidence of Adverse Events ≥ Grade 3 according to Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Incidence of TESAEs | 6 months
  Incidence of Related Treatment Emergent Serious Adverse Events (TESAEs) according to Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Overall Response Rate (ORR) by RECIST 1.1 | 6 months
  ORR is defined at Complete or Partial Response using local RECIST 1.1 compared to baseline
Overall Response Rate (ORR) by mRECIST | 6 months
  ORR is defined at Complete or Partial Response using local mRECIST compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — ABK Biomedical
Locations (1):
- Auckland District Health Board, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: No